CLINICAL TRIAL: NCT04788797
Title: Effect of the Endopeptidase AN-PEP on Gluten Exposure in Real Life in Celiac Disease Patients Treated With a Long-term Gluten-free Diet. Exploratory, Interventional, Prospective, Controlled and Double Blind Study
Brief Title: AN-PEP on Gluten Exposure in Celiacs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. C. Bonorino Udaondo Gastroenterology Hospital (Other Government)
Responsible Party: Principal Investigator, Edgardo Smecuol, Principal Investigator, Dr. C. Bonorino Udaondo Gastroenterology Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DrUdaondo
Record Dates: First submitted 2021-02-03; First posted 2021-03-09 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Celiac Disease
Keywords: celiac disease; endopeptidases; gliadin immunogenic peptides
MeSH Terms: conditions — Celiac Disease | interventions — Prolyl Oligopeptidases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prolyl Endopeptidase (Active Comparator): Patients blinded-receive active AN-PEP at a dose of 2 capsules/breakfast, lunch and dinner during 8 weeks (study arm)
  Interventions: Drug: Prolyl Endopeptidase
- Placebo (Placebo Comparator): Patients blinded-receive 2 capsules of a placebo (specially designed and prepared for the study) at breakfast, lunch and dinner during 8 weeks (Placebo arm).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prolyl Endopeptidase — Two capsules three times a day.
  Other Names: GliadinX
  Arms: Prolyl Endopeptidase
Other: Placebo — Two capsules three times a day
  Arms: Placebo

SUMMARY:
The AN-PEP, an Aspergillus niger derived endopeptidase, has been developed aiming to produce a complete luminal detoxification of gluten. If AN-PEP is able to produce a complete luminal digestion of gluten in the context of the real life of celiac disease (CeD) patients is unknown. Hypothetically, AN-PEP effect could be detected by the reduction in the excretion of GIP in stool and urine.

The objective of this study is to establish the effect of the daily administration of AN-PEP compared to placebo on GIP excretion in an interventional, prospective, randomized, comparative, double-blind study in conditions mimicking the real-life of CeD treated patients. The study consists in a four-week GFD stabilization period followed by a four-week study period with patients randomized to receive active AN-PEP or placebo in a blindly manner.

DETAILED DESCRIPTION:
Background: The strict gluten-free diet (GFD) is the only accepted treatment for celiac disease (CeD). However, performing a strict diet is still a non solved problem affecting the future of patients. In a real-life study it was recently shown that 89% of treated CeD patients performing a strict diet have contact with dietary gluten at least one week per 4 weeks of testing and averaging 3 weeks per month. Furthermore, 40% of patients excreted gliadin immunogenic peptides (GIP) (surrogated markers of gluten exposure) in the range for immunological activation and intestinal mucosal damage. Endopeptidases to produce a complete intraluminal proteolysis of gluten avoiding antigenic stimulation were produced to avoid damage of continuous gluten exposure. AN-PEP is an Aspergillus niger derived endopeptidase has been produced aiming to luminal detoxification of gluten have been explored for its clinical effect. However, whether AN-PEP is able to completely destroy gluten in the context of the real life of CeD patients is still unknown. Hypothesis: The investigators estimate that AN-PEP is an effective therapy for proteolysis for gluten exposure in the real-life of CeD patients and that the effect could be detected by the reduction in the excretion of GIP in stool and urine based on a clinical research model that we developed. AIMS: to establish the effect of daily administration of AN-PEP compared to placebo in terms of: (1) frequency of GIP excretion in stool and urine episodes in 4 weeks; (2) concentration of GIP excretion for both arms; and (3) differences in proportion of patients excreting GIP above the threshold for mucosal damage (>2 µg/g of GIP in stool or >12 ng/mL in urine). Study design: Interventional, prospective, randomized, comparative, double-blind study. Components: 1- four-week GFD stabilization period; 2-Randomization. 3- four4-week study period: Patients blinded-receive active AN-PEP (GliadinX®) at a dose of 2 capsules/breakfast, lunch and dinner (study arm), or 2 capsules at same time points of placebo (specially designed and prepared for the study) (Placebo arm).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Diagnosis of celiac disease
* Completion of Gluten-free Diet for at least two years without evidence of voluntary violations.
* Patients who do not report symptoms of constipation or illnesses or medications (cathartics, antidiarrheals, etc.) that alter the bowel movement rhythm (accepted rhythm: between 2 times / day to 1 every other day) and diuresis (diuretics). Proton-pump inhibitor.
* Signature of the informed consent

Exclusion Criteria:

* Patients not interested or unable to collaborate with the questionnaires and collection of fecal matter.
* Place of residence of the participant more than 4 hours from the hospital, which interferes with the viability of the sample.
* Complicated CD (refractory CD type II, ulcerative jejunoileitis, lymphoma).
* Concomitant pathologies that are decompensated or untreated at study entry (type I or II diabetes mellitus; hyperthyroidism; hypothyroidism; kidney failure,).

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of GIP excretion in stool | 4 weeks
  To establish the effect of daily administration of AN-PEP compared to placebo in terms of frequency of GIP excretion in stool episodes in 4 weeks.
Weekly concentration of GIP excretion in stool | 4 weeks
  To determine weekly concentration of GIP excretion in stool (µg/g of GIP) for both patients randomized to AN-PEP or placebo.
Proportion of patients excreting GIP | 4 weeks
  To establish the proportion of patients excreting GIP above the theoretical threshold for mucosal damage (>1.6 µg/g of GIP in stool or >12 ng/mL in urine)
Frequency of GIP excretion in urine | 4 weeks
  To establish the effect of daily administration of AN-PEP compared to placebo in terms of frequency of GIP excretion in urine epidodes in 4 weeks
Weekly concentration of GIP excretion in urine | 4 weeks
  To determine weekly concentration of GIP excretion in urine (ng/mL) for both patients randomized to AN-PEP or placebo.

SECONDARY OUTCOMES:
Clinical effect of AN-PEP vs placebo | 4 weeks
  2.1- To establish differences in the clinical effect of AN-PEP vs. placebo in symptomatic celiac patients in terms of the Celiac Clinical Score comparing baseline scores vs. those from the end of the study period. Celiac Clinical Score is made up of sixteen items, 11 of which evaluate "specific symptoms" and 5 evaluate "general health". Each question is answered on a Likert scale from 1 to 5. Overall symptom scores were calculated through simple addition, with higher scores denoting more severe symptoms. Scores of 45 or higher are associated with a relatively poor quality of life and worse GFD adherence. Score less than 45 are associated with better quality of life and gluten adherence
Differences in quality of life scores | 4 weeks
  To determine differences in quality of life according to the Short Form 36 questionnaire in the study period in symptomatic and asymptomatic patients. To score this questionnaire scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Major symptoms | 4 weeks
  To explore changes in the daily report of major symptoms (abdominal pain, discomfort, borborygmi, distension, diarrhea) (Likert scale of seven points) in symptomatic patients by using a daily report in a telephonic APP.
Biochemical effect of AN-PEP vs. placebo | 4 weeks
  to evaluate changes that occur during the study period in concentrations of CD-specific antibodies (IgA TG2 and DGP antibodies -AU/mL-) comparing consumption of AN-PEP vs. placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo G Smecuol, Study Chair — Dr. C. Bonorino Udaondo Gastroenterology Hospital
Locations (1):
- Dr. C. Bonorino Udaondo Gastroenterology Hospital, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinto-Sanchez MI, Hall GB, Ghajar K, Nardelli A, Bolino C, Lau JT, Martin FP, Cominetti O, Welsh C, Rieder A, Traynor J, Gregory C, De Palma G, Pigrau M, Ford AC, Macri J, Berger B, Bergonzelli G, Surette MG, Collins SM, Moayyedi P, Bercik P. Probiotic Bifidobacterium longum NCC3001 Reduces Depression Scores and Alters Brain Activity: A Pilot Study in Patients With Irritable Bowel Syndrome. Gastroenterology. 2017 Aug;153(2):448-459.e8. doi: 10.1053/j.gastro.2017.05.003. Epub 2017 May 5. PMID 28483500
- [Background] Castellano E, Attanasio R, Gianotti L, Cesario F, Tassone F, Borretta G. Forearm DXA Increases the Rate of Patients With Asymptomatic Primary Hyperparathyroidism Meeting Surgical Criteria. J Clin Endocrinol Metab. 2016 Jul;101(7):2728-32. doi: 10.1210/jc.2016-1513. Epub 2016 Apr 12. PMID 27070376
- [Background] Ricano-Ponce I, Gutierrez-Achury J, Costa AF, Deelen P, Kurilshikov A, Zorro MM, Platteel M, van der Graaf A; Consortium for the study of genetic associations of celiac disease in Latin-America; Sanna S, Daffra O, Zhernakova A, Fu J, Trynka G, Smecuol E, Niveloni SI, Bai JC, Kumar V, Wijmenga C. Immunochip meta-analysis in European and Argentinian populations identifies two novel genetic loci associated with celiac disease. Eur J Hum Genet. 2020 Mar;28(3):313-323. doi: 10.1038/s41431-019-0520-4. Epub 2019 Oct 7. PMID 31591516
- [Background] Pinto-Sanchez MI, Bai JC. Toward New Paradigms in the Follow Up of Adult Patients With Celiac Disease on a Gluten-Free Diet. Front Nutr. 2019 Oct 1;6:153. doi: 10.3389/fnut.2019.00153. eCollection 2019. PMID 31632977
- [Background] Penny HA, Raju SA, Lau MS, Marks LJ, Baggus EM, Bai JC, Bassotti G, Bontkes HJ, Carroccio A, Danciu M, Derakhshan MH, Ensari A, Ganji A, Green PHR, Johnson MW, Ishaq S, Lebwohl B, Levene A, Maxim R, Mohaghegh Shalmani H, Rostami-Nejad M, Rowlands D, Spiridon IA, Srivastava A, Volta U, Villanacci V, Wild G, Cross SS, Rostami K, Sanders DS. Accuracy of a no-biopsy approach for the diagnosis of coeliac disease across different adult cohorts. Gut. 2021 May;70(5):876-883. doi: 10.1136/gutjnl-2020-320913. Epub 2020 Nov 2. PMID 33139268
- [Background] Seiler CL, Kiflen M, Stefanolo JP, Bai JC, Bercik P, Kelly CP, Verdu EF, Moayyedi P, Pinto-Sanchez MI. Probiotics for Celiac Disease: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Gastroenterol. 2020 Oct;115(10):1584-1595. doi: 10.14309/ajg.0000000000000749. PMID 32740074
- [Background] Stefanolo JP, Talamo M, Dodds S, de la Paz Temprano M, Costa AF, Moreno ML, Pinto-Sanchez MI, Smecuol E, Vazquez H, Gonzalez A, Niveloni SI, Maurino E, Verdu EF, Bai JC. Real-World Gluten Exposure in Patients With Celiac Disease on Gluten-Free Diets, Determined From Gliadin Immunogenic Peptides in Urine and Fecal Samples. Clin Gastroenterol Hepatol. 2021 Mar;19(3):484-491.e1. doi: 10.1016/j.cgh.2020.03.038. Epub 2020 Mar 23. PMID 32217152
- [Background] Smecuol E, Constante M, Temprano MP, Costa AF, Moreno ML, Pinto-Sanchez MI, Vazquez H, Stefanolo JP, Gonzalez AF, D'Adamo CR, Niveloni SI, Maurino E, Verdu EF, Bai JC. Effect of Bifidobacterium infantis NLS super strain in symptomatic coeliac disease patients on long-term gluten-free diet - an exploratory study. Benef Microbes. 2020 Oct 12;11(6):527-534. doi: 10.3920/BM2020.0016. Epub 2020 Oct 9. PMID 33032471